CLINICAL TRIAL: NCT03551587
Title: Comparative Evaluation Of Postoperative Pain After Using Sonic Vibringe Irrigation System Versus Conventional Irrigation In Single Rooted Teeth With Symptomatic Irreversible Pulpitis : A Randomized Clinical Controlled Trial
Brief Title: Comparison Between the Vibringe and the Conventional Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara shehata, Postgraduate student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vibringe_Postoperative_pain
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Endodontic Inflammation
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigant delivered by the Vibringe (Experimental): Experimental group:
  The irrigant will be delivered and sonically activated with the Vibringe system.
  Interventions: Device: Vibringe
- Irrigation by Conventional needle (No Intervention): Control group:
  Irrigation procedures will br performed with a conventional method using conventional gauge 24 needle.

INTERVENTIONS:
Device: Vibringe — The Vibringe is the first endodontic sonic irrigation system that enables delivery and activation of the irrigation solution in the root canal, in only one step.
  Arms: Irrigant delivered by the Vibringe

SUMMARY:
The Vibringe is the first endodontic sonic irrigation system that enables delivery and activation of the irrigation solution in the root canal, in only one step. The activation of the disinfectant by acoustic streaming, enriches and completes the irrigation procedure and improves the success rate of endodontic treatments. It has been shown that this system significantly improves debridement. It also improves the disruption of the smear layer and biofilm by activating irrigation solutions.

As there are no previous studies comparing the Vibringe system with other irrigation techniques under clinical settings, in this regard, the aim of this study is to evaluate whether irrigation with Vibringe provides more or less benefit in terms of postoperative pain when compared with the conventional needle technique.

DETAILED DESCRIPTION:
Postoperative pain is defined as the sensation of discomfort after endodontic intervention and is reported by 25%-40% of patients irrespective of pulp and peri-radicular status. According to the 2011 systematic review of Pak and White , the prevalence of pain in the first 24 hours is 40%, falling to 11% after 7 days. Dentinal debris, pulp tissue, microorganisms and irrigants can be conveyed to the peri-radicular tissues during root canal preparation and such extrusion of debris can lead to postoperative complications, such as flare-ups.

Mechanical instrumentation and irrigation are used to remove vital and necrotic remnants of pulp tissue, debris, microbiota and their by-products from a root canal system. However, several studies using microcomputed tomography scanning imagery have shown that most of the areas of the main root canal wall remain untouched by the instruments. This emphasizes the importance of other means of cleaning and disinfecting all areas of the root canal.

To enhance the effectiveness of cleaning and disinfecting all areas of the root canal, several irrigants are commonly used as initial and final rinses to overcome the shortcomings of using a single irrigant, such as sodium hypochlorite (NaOCl), ethylene-diaminetetraacetic acid or chlorhexidine. In addition to these various irrigants, numerous irrigation devices and needle tips have been developed with the aim of improving the delivery of irrigant throughout the root canal using sonic or ultrasonic energy and negative apical pressure.

However, as well as the success of the irrigation devices in removing debris from the root canal, a safe irrigation delivery system is desirable to prevent periapical tissue damage and decrease post-endodontic pain. The available data on extrusion of irrigant when using these devices appears to be limited to laboratory studies.

Rationale :

The Vibringe is the first endodontic sonic irrigation system that enables delivery and activation of the irrigation solution in the root canal, in only one step. The activation of the disinfectant by acoustic streaming, enriches and completes the irrigation procedure and improves the success rate of endodontic treatments. It has been shown that this system significantly improves debridement. It also improves the disruption of the smear layer and biofilm by activating irrigation solutions.

Vasconcelos et al at in vitro study at 2017 proved that groups using ultrasonic agitation presented a greater antibacterial effect than the other ones, even using saline solution as irrigant. Middha et al studied the effect of continuous ultrasonic irrigation on postoperative pain in mandibular molars with nonvital pulps concluded that a significant difference was observed between CUI and syringe irrigation on the first postoperative day following chemo-mechanical preparation. However, the benefit observed was not clinically relevant.

It has been shown that the Vibringe results in an equal performance in canal and isthmus debridement efficacy when compared with needle irrigation in the apical region (9). In addition, it did not significantly alter sealer penetration compared with conventional needles. Furthermore, another recent study concluded that the Vibringe extruded more debris than conventional needle irrigation .

Postoperative pain associated with root canal treatment is a poor indicator of long-term success; however, the occurrence and the control of pain are of clinical interest. So , this study will focus on evaluating postoperative discomfort due to the fact that Vibringe is an actively vibrating system, which may lead to postoperative discomfort.

Objective of the study :

As there are no previous studies comparing the Vibringe system with other irrigation techniques under clinical settings, in this regard, the aim of this study is to evaluate whether irrigation with Vibringe provides more or less benefit in terms of postoperative pain when compared with the conventional needle technique.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-45 years old.
* Males or Females.
* Single rooted teeth with:
* Symptomatic irreversible pulpitis .
* Normal periapical radiographic appearance or slight widening in lamina dura.

Exclusion Criteria:

* Patients on medication for chronic pain.
* Patients having significant systemic disorders.
* Teeth that have :
* Vital pulp tissues.
* Swelling or fistulous tract
* Acute or chronic peri-apical abscess
* Greater than grade I mobility
* Pocket depth greater than 5mm
* No possible restorability
* Previous endodontic treatment.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-01-27 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
pain intensity ( post operative pain ) | 6 hours post- obturation.
  post operative pain measured by Numeric Rating Scale (0-10) where; 0; No pain. 1-3; Mild Pain 4-6; Moderate Pain 7-10; Severe pain: "severe pain, analgesic had no effect in relieving the pain".
pain intensity ( post operative pain ) | 12 hours post- obturation.
  post operative pain measured by Numeric Rating Scale (0-10) where; 0; No pain. 1-3; Mild Pain 4-6; Moderate Pain 7-10; Severe pain: "severe pain, analgesic had no effect in relieving the pain".
pain intensity ( post operative pain ) | 24 hours post- obturation.
  post operative pain measured by Numeric Rating Scale (0-10) where; 0; No pain. 1-3; Mild Pain 4-6; Moderate Pain 7-10; Severe pain: "severe pain, analgesic had no effect in relieving the pain".
pain intensity ( post operative pain ) | 48 hours post- obturation.
  post operative pain measured by Numeric Rating Scale (0-10) where; 0; No pain. 1-3; Mild Pain 4-6; Moderate Pain 7-10; Severe pain: "severe pain, analgesic had no effect in relieving the pain".

CONTACTS AND LOCATIONS:
Overall Officials: Professor Heba El Far, Study Director — Cairo University; Faculty of Dentistry, Study Chair — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt